## COMPLUTENSE UNIVERSITY OF MADRID FACULTY OF NURSING, PHYSIOTHERAPY AND PODIATRY



## TITLE: CLINICAL TRIAL WITHOUT MEDICATION: PREVENTION OF BODY IMAGE DISORDER FOR NURSING INTERVENTION ON PATIENT AND FAMILY PRIOR TO MAMA AND COLON CANCER SURGERY

## MEMORY TO CHOOSE THE DEGREE OF DOCTOR PRESENTED BY

Natalia Mudarra García

Under the direction of the doctors

Enrique Pacheco Del Cerro Alfonso Meneses Morroy

Madrid, 2018

## INFORMED CONSENT FORM

I confirm that I have read the information sheet about the study mentioned above, I have received enough information about the study and that I have had the opportunity to ask questions.

I understand that my participation is voluntary and that I am free to leave the study at any time, without giving any explanation and without my medical care or legal rights being affected by this circumstance.

I freely give my consent to participate in the study and give my consent for the access and use of my data in the conditions detailed in the information sheet.

I give permission for these people to have access to my medical record.

I agree to participate in the aforementioned study.

I can make use of the rights of L.O. 15/1999 of Protection of Personal Data.

Sign the copy of the informed consent for the researcher and the copy for the participant.

Name / family of the relative who will accompany you in the study.